CLINICAL TRIAL: NCT02430103
Title: Effect of Goserelin on the Protection of Ovarian Reserve During (Neo)Adjuvant Chemotherapy for Young Breast Cancer Patients: A Prospective Cohort Trial
Brief Title: Study of Preservation of Ovarian Reserve During Chemotherapy for Young Breast Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Siyuan Wang, Nothing, Peking University People's Hospital
Other Study IDs: PKUPHBC-001
Record Dates: First submitted 2015-04-06; First posted 2015-04-30 (Estimated); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Preservation of Ovarian Reserve Function; Goserelin; AMH
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (2):
- Chemotherapy plus GnRHa: Patients of the group will receive (neo)chemotherapy plus GnRHa ( Goserelin 3.6mg will be administered every 28 days by subcutaneous injection starting at least 7-14 days before the first cycle of chemotherapy and continued throughout chemotherapy duration).
  Interventions: Drug: Goserelin 3.6 MG
- Chemotherapy: Patients of the group will receive (neo)chemotherapy merely.

INTERVENTIONS:
Drug: Goserelin 3.6 MG — In goserelin group, goserelin 3.6mg will be administered every 28 days by subcutaneous injection starting at least 7-14 days before the first cycle of chemotherapy and continued throughout chemotherapy duration.
  Other Names: Zoladex
  Groups: Chemotherapy plus GnRHa

SUMMARY:
The purpose of this study is to assess efficacy of gonadotropin-releasing hormone agonist (goserelin) on the preservation of ovarian reserve function in young breast cancer patients treated with (neo)adjuvant chemotherapy by serial measuring ovarian reserve markers (AMH and AFC.etc) before and after chemotherapy and long-term pregnancy outcomes. Meanwhile, to evaluate the safety of this protective approach in young breast cancer patients by disease-free survival (DFS) and overall survival (OS) outcomes.

DETAILED DESCRIPTION:
6.6-12% of women with breast cancer were diagnosed before the age of 40 year and breast cancer accounted for 40% of all cancer in women before the age of 40 year.Attributed to improved treatment, of which chemotherapy plays a major role, more than 70% of breast cancer patients at reproductive age obtain 10-year survival rates. Consequently, the question of pregnancy and premature ovarian failure after breast cancer treatment are presented more frequently. Fortunately, most of the available literature provides good evidence that pregnancy after breast cancer may improve survival. Unfortunately, no therapy has been shown to preserve fertility in patients receiving chemotherapy so far, although chemotherapy induced ovarian failure ,which finally results in infertility and premature ovarian failure, has been reported 60 years before. The greater rate of prepubertal than of postpubertal women with normal ovarian function after chemotherapy supports the concept that the suppressed ovary has a greater tolerance during cytotoxic treatments.While inhibiting the pituitary ovarian axis, Gonadotropin-releasing hormone agonist (GnRHa) is thought to block follicular development and reduce chemotherapy toxicity. Several studies had revealed GnRHa co-treatment yielded a statistically significant improvement in the proportion of spontaneous menstrual resumption after chemotherapy, compared to controls.It is noteworthy that menses and fertility are not necessarily linked. Absence of regular menses, particularly if the patient is taking tamoxifen(endocrine therapy for breast cancer), does not necessarily imply lack of fertility. Conversely, the presence of menses does not guarantee fertility.Currently, anti-Müllerian hormone(AMH) is considered as the best biochemical marker for assessment of reproductive capacity in reproductive medicine settings. Because it is produced by granulosa cells of growing antral follicles, AMH is significant positive correlation with both quantity and quality of oocytes. Moreover, it can be measured on any day for minimal fluctuation during the menstrual cycle.Antral follicle count (AFC) by vaginal ultrasound is also a good predictor of response to exogenous FSH and correlates independently with the number of oocytes retrieved during in vitro fertilization(IVF). Our study is designed to make sure the effect of GnRHa on the preservation of ovarian reserve function in breast cancer patients at reproductive age treated with (neo)adjuvant chemotherapy by observing the dynamic changes of ovarian reserve marker (AMH, AFC, E2 and FSH) pre and post chemotherapy and long-term pregnancy outcomes. Meanwhile, to evaluate the safety of this protective approach in young breast cancer patients by disease-free survival (DFS) and overall survival (OS) outcomes, and objective response rate(ORR) and pathological complete response (pCR) rate (for patitents treated with neoadjuvant chemotherapy). Finally, to explore whether patients with GnRH receptor or androgen receptor over-expression could benefit survival from this approach.

Patients: Premenopausal patients aged 18-45 years were eligible for enrollment, with stages I to III of newly diagnosed breast cancer, for which treatment with adjuvant or neoadjuvant chemotherapy was planned. Exceptions were made up of the use of hormonal contraception, previous chemotherapy, bilateral oophorectomy or ovarian irradiation before enrollment, and GnRHa -containing endocrine therapy planned.

Study Design: In our study, patients will be informed comprehensively and assigned without interference to receive either (neo)adjuvant chemotherapy with goserelin (goserelin group) or without goserelin (chemotherapy group) as their own selection. AMH, follicle stimulating hormone (FSH), and estradiol (E2) are used as biochemical markers and AFC is used as biophysical marker. The markers and menstrual status will be evaluated before, during, and at 0.5-year, 1-year, 2-year after chemotherapy. Additionally, pregnancy and disease related outcomes within 5 years, assessed annually.

Patients in goserelin group are given a subcutaneously dose of 3.6 mg (Zoladex, AstraZeneca) at least 1 week before the first cycle of chemotherapy and then every 4 weeks for the duration of chemotherapy. Subgroup analysis is stratified by age (≤ 40 years and 41-45 years), baseline level of AMH(≤1ng/ml and >1ng/ml), chemotherapy regimen (AC, AC-T(H), others) and endocrine therapy regimen (with or without Tamoxifen).

The primary end point is to compare the recovery rate of AMH value (≥ 0.5ng/ml) (according to the "the Bologna criteria") between the two treatment groups at 2-year after chemotherapy. Secondary endpoints included descriptions of the dynamic changes of each marker from pre- to post-chemotherapy and time to resumption of menstrual activity (reappearance of two consecutive menstrual periods within 21 to 35 days); recovery rate of AMH value at 1 year and the rates of the other markers returning to the premenopausal range (E2 ≥ 40 pg/ml, FSH < 25 U/L, AFC ≥ 5) were assessed at both 1 year and 2 years. Additional end points included pregnancy and disease related outcomes within 5 years, assessed annually. Events in the analysis of disease-free survival (DFS) included local recurrence, distant metastases, contralateral or ipsilateral breast tumor, second primary malignancy, and death due to any cause. Events in the analysis of overall survival (OS) included deaths due to any cause. Explore whether patients with GnRH receptor or androgen receptor over-expression could benefit survival by subtype analysis.

Statistical Analysis: Sample size calculation was based on the GBG 37 ZORO study. Out of 60 patients, 17 were accessible for AMH assessment during follow up to estimate ovarian function in 24 months after end of chemotherapy. Out of these 17 patients, 8 received goserelin and 9 were treated without goserelin. Recovery to normal AMH level was seen in 3 of 9 (33%) patients in chemotherapy group vs 4 of 8 (50%) patients in goserelin group respectively. To have 80% power to detect a 17% improvement in recovery to normal AMH level in 2 years, with a two-sided type I error rate of 0.05, 230 patients were needed to be assigned (calculated by NCSS-PASS). Finally, considering dropping off of patients, the target enrollment was 240 eligible patients. Descriptive statistics of baseline demographics and clinicopathologic characteristics were considered in the two treatment groups.The recovery rates of ovarian reserve markers and menses at 1-year and 2-year follow-up after chemotherapy were compared by a Pearson chi-square test. Logistic regression was performed to study the effect of age, baseline level of AMH, chemotherapy regimen and tamoxifen possible interactions on the probability of ovarian recovery. The differences in the baseline clinicopathological characteristics between the two groups were adjusted through propensity score weighting. The propensity score for each patient was estimated by a logistic regression model using group (the chemotherapy group or the goserelin group) as dependent variable and all patient characteristics as independent variables. Next, adjusted recovery rates of these markers and menses were compared by the chi-square test. Hormone concentrations and AFC at each time point were compared using the Mann-Whitney test. Log-rank statistics was used to compare time to return of menses between the two groups. Finally, Kaplan-Meier curve for disease-free will be calculated and compared by log-rank test. P values less than 0.05 are considered statistically significant. Analyses are performed by using SPSS version 18 software.

In summary: our study is the first prospective cohort study that focus on the premenopausal breast cancer patients who would like to preserve the ovarian function in China. The results will be more adaptable in China and other countries in Asia where breast cancer patients' age at diagnosis is younger. The outcome of this study may offer breast cancer patients at reproductive age hope of becoming mothers and possessing vigour of youth.

Recent breast cancer treatment guidelines strongly recommended that moderate and high-risk young patients with hormone receptor-positive disease should receive ovarian function suppression as part of adjuvant endocrine therapy, based largely on the results of the SOFT and TEXT Trials. Consequently, more than 20% patients in the two treatment group in this study who had hormone receptor-positive disease were estimated to directly receive or to change from tamoxifen to a GnRHa-containing endocrine therapy regimen and would not be assessed at the 2-year follow-up after chemotherapy. Therefore, an interim statistical analysis was determined to perform on the eligible patients who could be evaluated at 1 year after chemotherapy in the two treatment groups. The cutoff date for this analysis was November 30, 2019.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients must fulfil all of the following criteria:

1. Aged 45 years or younger
2. Have regular menstrual cycle
3. Newly diagnosed early-stage breast cancer (stages I to III)
4. Planned (neo)adjuvant chemotherapy
5. Signed informed consent document on file

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Pregnancy or lactation
2. Oral contraceptives before enrollment
3. Prior chemotherapy
4. Bilateral oophorectomy or ovarian irradiation before enrollment
5. History of other cancers
6. GnRHa -containing adjuvant endocrine therapy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 240 premenopausal breast cancer patients of age 45 years or younger treated in Peking University People's Hospital Breast Center
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2015-12-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery of serum AMH value(≥0.5ng/ml) in 2 years of post-chemotherapy | Phlebotomy will be carried out at 2 years (one month ahead or one month delayed could be accepted) after chemotherapy in both groups.
  AMH can be measured on any day during the menstrual cycle.Serum AMH concentrations will be measured using the AMH Gen II ELISA, according to the manufacturer's instructions

SECONDARY OUTCOMES:
Recovery of AFC (≥5) by ultrasound per vagina in 1 year and 2 years of post-chemotherapy | AFC will be performed at 1 year and 2 years (one month ahead or one month delayed could be accepted) after chemotherapy in both groups.
  AFC by ultrasound per vagina will be performed by the physician from Peking University People's Hospital Reproductive Medicine Center. AFC for virginity will be performed by ultrasound per rectum. The optimal date of measuring AFC is the days after menstruation.

OTHER OUTCOMES:
Recovery of serum Follicle-Stimulating Hormone (FSH<25U/L) in 1 year and 2 years of post-chemotherapy | Phlebotomy will be carried out at 1 year and 2 years (one month ahead or one month delayed could be accepted) after chemotherapy in both groups.
  When menses are regular, the optimal date of phlebotomy is on day 2-5 during the cycle.
Recovery of serum Estradiol (E2≥40pg/ml) in 1 year and 2 years of post-chemotherapy | Phlebotomy will be carried out at 1 year and 2 years (one month ahead or one month delayed could be accepted) after chemotherapy in both groups.
  When menses are regular, the optimal date of phlebotomy is on day 2-5 during the cycle.
Recovery of serum AMH value(≥0.5ng/ml) in 1 year of post-chemotherapy | Phlebotomy will be carried out at 1 year (one month ahead or one month delayed could be accepted) after chemotherapy in both groups.
  AMH can be measured on any day during the menstrual cycle.Serum AMH concentrations will be measured using the AMH Gen II ELISA, according to the manufacturer's instructions
Resumed menses in 1 year and 2 years of post-chemotherapy | Evaluation of menses at 1 year and 2 years after chemotherapy in both groups.
  reappearance of two consecutive menstrual periods within 21 to 35 days after chemotherapy
Disease-free survival | Evaluation of disease-free survival annually after chemotherapy in both groups.
  Events in the analysis of disease-free survival include local recurrence, distant metastases, contralateral or ipsilateral breast tumor, second primary malignancy, and death due to any cause.
Overall survival | Evaluation of overall survival annually after chemotherapy in both groups.
  Events in the analysis of overall survival included deaths due to any cause.
Pregnancy | Pregnancy outcome assessed annually after chemotherapy in both groups.
  Pregnancy event after chemotherapy in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, Principal Investigator — Peking University People's Hospital Breast Center
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Wang S, Pei L, Hu T, Jia M, Wang S. Protective effect of goserelin on ovarian reserve during (neo)adjuvant chemotherapy in young breast cancer patients: a prospective cohort study in China. Hum Reprod. 2021 Mar 18;36(4):976-986. doi: 10.1093/humrep/deaa349. PMID 33411897